CLINICAL TRIAL: NCT03300869
Title: Natural History of Types 2 and 3 Spinal Muscular Atrophy in Taiwan
Brief Title: Natural History of Types 2 and 3 SMA in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Biogen (Industry); National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); China Medical University Hospital (Other); Changhua Christian Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMA_RV
Record Dates: First submitted 2017-09-13; First posted 2017-10-04 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Natural History
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to investigate the natural history of spinal muscular atrophy (SMA) types 2 and 3 patients in Taiwan. This study will provide further insights into the clinical course SMA. Several analyses will be conducted regarding overall survival, demographic characteristics, motor function, respiratory and nutritional support, and genotype and phenotype correlation.

DETAILED DESCRIPTION:
As with other rare diseases, individual groups of SMA have therefore opted to share patient information in the form of clinical sites to increase the overall patient cohorts on which clinical outcomes and new assisted-healthcare technologies can be assessed. Using the collaborative and retrospective study of types 2 and 3 SMA patients in Taiwan, the investigators aim to 1) characterize the correlation of genotype and phenotype, 2) correlate the onset, progression, management with disease outcome, 3) depict comorbidity and within type 2 and 3 SMA patients with different SMN2 copy number.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are diagnosed with SMA types 2 or 3
2. Generalized hypotonia and muscle weakness, weakness of the legs is greater than the arms, and the proximal part is weaker than distal part of extremities.
3. SMN1 gene deletion or mutation and/or neurogenic changes in electromyogram and/or muscle pathology.

Exclusion Criteria:

1. Non-5q SMA (no deletion or mutation of SMN1 gene) patients.
2. Type 1 SMA patients.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the past decades, The SMA is a rare disease (incidence of 1 in every 6,000-10,000 live births) with a carrier frequency of about 1 in 40-50 people. Therefore, individual countries have small cohorts of affected patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Describe the correlation of genotype and phenotype in SMA types 2 and 3 | through study completion, an average of 2 years
  Genotype is defined by SMN 2 copy number(s) and phenotype is defined by clinical types and characteristics.

SECONDARY OUTCOMES:
Disease onset in patients with SMA types 2 and 3 | through study completion, an average of 2 years
  Number of participants with disease onset as assessed by year
Disease mortality in patients with SMA types 2 and 3 | through study completion, an average of 2 years
  Number of participants with disease mortality as assessed by year
Scoliosis in patients with SMA types 2 and 3 | through study completion, an average of 2 years
  Number of participants with scoliosis as assessed by year
BiPAP usage in patients with SMA types 2 and 3 | through study completion, an average of 2 years
  Number of participants with BiPAP usage as assessed by year

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available